CLINICAL TRIAL: NCT00732355
Title: One-Step Syphilis Point of Care Test for Rapid Immunoassay Screening of Antibodies to Treponema Pallidum
Brief Title: Syph-Check Syphilis Antibody Point of Care (POC) Test
Acronym: SyphPoc
Status: Terminated | Type: Observational
Why Stopped: insufficient patient populations
Sponsor: Healthcare Providers Direct, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SY-101
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Screening for Syphilis Infections
Keywords: syphilis
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- I: known syphilis infected patients
  Interventions: Device: Syph-Check POC
- U: presumed uninfected patients
  Interventions: Device: Syph-Check POC

INTERVENTIONS:
Device: Syph-Check POC — Rapid membrane test for syphilis antibodies
  Other Names: RPR; TPPA; syphilis

SUMMARY:
The study is designed to evaluate the performance of a rapid membrane test in a clinic or doctor's office setting to identify potential patients infected with syphilis and compare the results to currently licensed laboratory based tests.

DETAILED DESCRIPTION:
The overall objectives of this study are to determine the performance characteristics of a candidate rapid point-of-care test (Syph-Check cassette format) for Treponema pallidum antibodies in serum, plasma and finger stick whole blood obtained from females and males attending sexually transmitted diseases (STD) clinics, family planning / reproductive health clinics, and physician's office; and to compare the performance of this new, rapid test to currently licensed laboratory based tests, the non-treponemal RPR and a Treponemal ELISA or TPPA test.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women will be eligible who:

  1. are 18 years of age or older;
  2. Routine "presumed uninfected" for screening visit, or show symptomatic signs of infection or are asymptomatic but are suspected of infection, and either/or have other STD disease conditions and infections, will be identified.
  3. Pregnant women in the first and third trimester

Exclusion Criteria:

* are under 18 years of age
* unwillingness to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Point of Care clinics and doctor's office that test routine patients (both male and female), i.e. STD clinics, planned parenthood, pre-marital, blood donors, pre-employment, and general populations from different geographic locations having varying prevalence populations.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Identify the sensitivity and specificity of the POC test versus accepted laboratory tests | end of study

SECONDARY OUTCOMES:
Percent positive agreement data will include supplemental test results identified by infection categories and treatment as possible | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Gary L Lehnus, Ph.D., Study Director — Lehnus & Associates Consulting
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No